CLINICAL TRIAL: NCT00381342
Title: Safety and Efficacy of Exenatide as Monotherapy in Drug Naive Patients With Type 2 Diabetes
Brief Title: Safety and Efficacy of Exenatide as Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-MC-GWBJ
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; Amylin; Lilly; monotherapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exenatide 5 mcg/exenatide 5 mcg (Experimental): Exenatide 5 mcg; then exenatide 5 mcg
  Interventions: Drug: exenatide
- Exenatide 5 mcg/exenatide 10 mcg (Experimental): Exenatide 5 mcg, then exenatide 10 mcg
  Interventions: Drug: exenatide
- Placebo (Placebo Comparator): Placebo in volumes equivalent to exenatide
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: exenatide — Placebo subcutaneously injected twice daily as a lead-in followed by exenatide subcutaneously injected, 5 mcg, twice a day
  Other Names: Byetta
  Arms: Exenatide 5 mcg/exenatide 5 mcg
Drug: exenatide — Placebo subcutaneously injected twice daily as a lead-in followed by exenatide subcutaneously injected, 5 mcg, twice a day, then exenatide subcutaneous injection, 10 mcg twice a day
  Other Names: Byetta
  Arms: Exenatide 5 mcg/exenatide 10 mcg
Drug: placebo — subcutaneous injection, volume equivalent to appropriate dose of exenatide, twice a day
  Arms: Placebo

SUMMARY:
This Phase 3 trial is designed to compare the effects of twice-daily exenatide and twice-daily placebo with respect to glycemic control in drug-naive patients with type 2 diabetes treated with diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Treating diabetes with diet and exercise
* HbA1c between 6.5% and 10.0%, inclusive
* Body Mass Index (BMI) between 25 kg/m^2 and 45 kg/m^2, inclusive

Exclusion Criteria:

* Have previously completed or withdrawn from this study
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Have been treated with any antidiabetic agent
* Have used drugs for weight loss (for example, Xenical, Meridia, Acutrim, or similar over-the counter medications) within 3 months of screening
* Are currently treated with any of the following excluded medications: * drugs that directly affect gastrointestinal motility; * systemic corticosteroids (excluding topical and inhaled preparations) by oral, intravenous, or intramuscular route used regularly (longer than 2 weeks) or used within 2 weeks immediately prior to screening for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated hemoglobin) from Baseline to Week 24 | Baseline, Week 24
  Change in HbA1c from Baseline to Week 24

SECONDARY OUTCOMES:
Percentage of subjects achieving HbA1c of 7% or less and of 6.5% or less | Baseline, Weeks 4, 8, 12, 16, 24
  Percentage of subjects achieving HbA1c of 7% or less and of 6.5% or less
Change in fasting serum glucose (FSG) from Baseline to Week 24 | Baseline, Weeks 4, 8, 12, 16, and 24
  Change in fasting serum glucose (FSG) from Baseline to Week 24 and, if measured, at all visits in between
Change in body weight from Baseline to Week 24 | Baseline, Weeks 4, 8, 12, 16, and 24
  Change in body weight (kg) from Baseline to Week 24 and, if measured, at all visits in between
Change in glucose measurements from Baseline to Week 24 | Baseline, Weeks 4, 8, 12, 16, 24
  Change in fasting SMBG profiles (glucose measurements before and 2 hours after meals) from Baseline to Week 24 and, if measured, at all visits in between
Changes in beta-cell function and insulin sensitivity from Baseline to Week 24 | Baseline, Weeks 4, 8, 12, 16, and 24
  Changes in beta-cell function and insulin sensitivity as assessed by homeostasis model assessment (HOMA) analyses from Baseline to Week 24 and, if measured, at all visits in between
Changes in fasting and 30, 60, 120 and 180-minute glucose measurements | Immediately before glucose load, then 30, 60, 120, and 180 minutes post
  Changes in fasting and 30, 60, 120, 180-minute post glucose load blood concentrations of glucose and insulin

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (19):
- United States (2):
  - Research Site, Idaho Falls, Idaho
  - Research Site, Indianapolis, Indiana
- India (7):
  - Research Site, Aligarh
  - Research Site, Bangalore
  - Research Site, Chennai
  - Research Site, Indore
  - Research Site, Karnāl
  - Research Site, New Delhi
  - Research Site, Vellore
- Puerto Rico (2):
  - Research Site, Manatí
  - Research Site, San Juan
- Romania (6):
  - Research Site, Alba Iulia
  - Research Site, Baia Mare
  - Research Site, Bucharest
  - Research Site, Galati
  - Research Site, Oradea
  - Research Site, Târgu Mureş
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg

REFERENCES:
- [Result] Moretto TJ, Milton DR, Ridge TD, Macconell LA, Okerson T, Wolka AM, Brodows RG. Efficacy and tolerability of exenatide monotherapy over 24 weeks in antidiabetic drug-naive patients with type 2 diabetes: a randomized, double-blind, placebo-controlled, parallel-group study. Clin Ther. 2008 Aug;30(8):1448-60. doi: 10.1016/j.clinthera.2008.08.006. PMID 18803987
- [Derived] Pencek R, Blickensderfer A, Li Y, Brunell SC, Anderson PW. Exenatide twice daily: analysis of effectiveness and safety data stratified by age, sex, race, duration of diabetes, and body mass index. Postgrad Med. 2012 Jul;124(4):21-32. doi: 10.3810/pgm.2012.07.2567. PMID 22913891
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356